CLINICAL TRIAL: NCT04523363
Title: Metformin Versus Standard of Care Treatment in Pregnant Women With Prediabetes: A Randomized Trial
Brief Title: Metformin Versus Standard of Care Treatment in Pregnant Women With Prediabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not funded and could not be performed
Sponsor: Gianna Wilkie (Other)
Responsible Party: Sponsor-Investigator, Gianna Wilkie, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00021261
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Prediabetes; Complicating Pregnancy
Keywords: maternal outcomes; neonatal outcomes; metformin; prediabetes; pregnancy
MeSH Terms: conditions — Prediabetic State; Pregnancy Complications | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This is a prospective, single center, randomized study evaluating metformin in the treatment of pregnant women with prediabetes on maternal and neonatal outcomes.
Who Masked: Outcomes Assessor
Masking Description: Those assessing the outcomes from the medical chart will be blinded to the randomization process and the assigned study arm. Patients, the primary investigator, and their care providers will be aware of their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Study subjects will be randomized to the metformin medication arm. They will take a 500 mg tablet orally twice a day starting at 14 weeks of pregnancy until delivery.
  Interventions: Drug: Metformin
- Standard of Care (No Intervention): Study subjects will be randomized to standard of care and receive routine prenatal care without further intervention for their prediabetes.

INTERVENTIONS:
Drug: Metformin — Maximum dosage of 500 mg tablets 2 times a day (with each meal)
  Other Names: Glucophage
  Arms: Metformin

SUMMARY:
The purpose of this study is to assess if metformin reduces adverse outcomes associated with prediabetes in pregnancy. Our hypothesis is that pregnant women with prediabetes who are treated with metformin will show a greater reduction in large for gestational age infants at birth compared to women treated with the standard of care.

DETAILED DESCRIPTION:
Women in pregnancy are routinely screened for diabetes in the first trimester and those who fall into the prediabetes category by hemoglobin A1c level of 5.7 to 6.4%, fasting plasma glucose of greater than or equal to 100 to 125, or oral glucose tolerance test of greater than or equal to 140 to less than 200 before 14 weeks gestation will be approached for consent in our randomized trial.

Once consent is obtained, the subjects will be randomized 1:1 into two parallel groups, the metformin treatment group and the standard of care treatment group (routine prenatal care). A random number generator will allocate the participants to the study groups.

Women taking metformin will continue twice daily dosing for the duration of their pregnancy after randomization. Those in the standard of care group will receive routine prenatal care. Both groups will undergo routine gestational diabetes testing by 28 weeks. Obstetric, maternal, and neonatal outcomes will then be assessed of both groups until the 6 week postpartum visit.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with hemoglobin A1c of 5.7 to 6.4%, fasting plasma glucose of greater than or equal to 100 to 125, or oral glucose tolerance test of greater than or equal to 140 to less than 200 before 14 weeks gestation
* Pregnancy and delivery care obtained at University of Massachusetts (UMass) Memorial Medical Center
* Patients able to provide written informed consent

Exclusion Criteria:

* Pre-existing diabetes diagnosis as assessed at visit in the first trimester by history or by laboratory evaluation as listed above
* Presence of contra-indication to metformin (liver, renal, or heart failure) or sensitivity to metformin
* Participants who are under the age of 18
* Multiple Pregnancy
* Patients already taking metformin for other indications
* Fetal defect noted on early dating ultrasound
* Miscarriage before randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Birth Weight | At Birth
  Used to determine large for gestational age status

SECONDARY OUTCOMES:
Number of Participants needing Cesarean Section | At Delivery
  Number of Participants with Cesarean Section
Number of Participants with Postpartum Hemorrhage | At Delivery
  Estimated or quantitative blood loss greater than 1000 mL
Number of Participants with Development of Pregnancy Induced Hypertension | Through study completion, starting at 14 weeks until delivery
  Blood pressure, serum laboratory analysis, and urine protein would be assessed for diagnosis
Development of Gestational Diabetes | Assessed at 28 weeks of pregnancy
  A glucose tolerance test would be conducted at 28 weeks of pregnancy to diagnose diabetes
Maternal Weight Gain in Pregnancy | At enrollment and last prenatal visit, starting at 14 weeks until delivery
Pregnancy Outcome | Through study completion, starting at 14 weeks until delivery
  Number of Participants with Stillbirth, livebirth, pregnancy loss
Number of Participants with Preterm birth | At delivery
  Less than 37 week delivery
Neonatal Intensive Care Unit Admission | At delivery and within first 2 days of life
  Admission to level 2 or greater neonatal ICU and length of stay
Apgar Score at Birth | At delivery
  <6 at 1 and 5 minutes
Number of Participants with Neonatal Birth Trauma | At Delivery
  Brachial plexus injury
Number of Participants with Shoulder Dystocia | At Delivery
Number of Participants with Neonatal Hypoglycemia | Within first 2 days of life
Number of Participants with Neonatal Respiratory Distress | At Delivery
  Requiring 2 or more hours of respiratory support or oxygen with associated diagnosis
Number of Participants with Neonatal Hyperbilirubinemia | Within first 2 days of life
  Requiring phototherapy
Number of Participants requiring Neonatal Intubation | At Delivery
Neonatal Cooling | Within first 2 days of life
  Need for neonatal cooling within first 48 hours of life
Umbilical Cord Blood Level of C-peptide | At Birth
Umbilical Cord Blood Level of Leptin | At Birth
Umbilical Cord Blood Level of Insulin | At Birth
Placental Pathology | At Birth
  Assessing for malperfusion pathology

CONTACTS AND LOCATIONS:
Overall Officials: Gianna L Wilkie, MD, Principal Investigator — UMass Memorial Health
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson C, Grosse SD, Li R, Sharma AJ, Razzaghi H, Herman WH, Gilboa SM. Preventable health and cost burden of adverse birth outcomes associated with pregestational diabetes in the United States. Am J Obstet Gynecol. 2015 Jan;212(1):74.e1-9. doi: 10.1016/j.ajog.2014.09.009. Epub 2014 Oct 28. PMID 25439811
- [Background] Lawrence JM, Contreras R, Chen W, Sacks DA. Trends in the prevalence of preexisting diabetes and gestational diabetes mellitus among a racially/ethnically diverse population of pregnant women, 1999-2005. Diabetes Care. 2008 May;31(5):899-904. doi: 10.2337/dc07-2345. Epub 2008 Jan 25. PMID 18223030
- [Background] Temple R, Murphy H. Type 2 diabetes in pregnancy - An increasing problem. Best Pract Res Clin Endocrinol Metab. 2010 Aug;24(4):591-603. doi: 10.1016/j.beem.2010.05.011. PMID 20832738
- [Background] Lee AM, Fermin CR, Filipp SL, Gurka MJ, DeBoer MD. Examining trends in prediabetes and its relationship with the metabolic syndrome in US adolescents, 1999-2014. Acta Diabetol. 2017 Apr;54(4):373-381. doi: 10.1007/s00592-016-0958-6. Epub 2017 Jan 9. PMID 28070750
- [Background] Chen L, Pocobelli G, Yu O, Shortreed SM, Osmundson SS, Fuller S, Wartko PD, Mcculloch D, Warwick S, Newton KM, Dublin S. Early Pregnancy Hemoglobin A1C and Pregnancy Outcomes: A Population-Based Study. Am J Perinatol. 2019 Aug;36(10):1045-1053. doi: 10.1055/s-0038-1675619. Epub 2018 Nov 30. PMID 30500961
- [Background] Professional Practice Committee for the Standards of Medical Care in Diabetes-2016. Diabetes Care. 2016 Jan;39 Suppl 1:S107-8. doi: 10.2337/dc16-S018. No abstract available. PMID 26696673